CLINICAL TRIAL: NCT04329117
Title: Society for Pediatric Anesthesia Improvement Network- Anterior Cruciate Ligament Reconstruction Outcomes Project
Acronym: SPAIN-ACL
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); Johns Hopkins University (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital Los Angeles (Other); University of Texas Southwestern Medical Center (Other); Duke University (Other); Alfred I. duPont Hospital for Children (Other); Akron Children's Hospital (Other); Children's National Research Institute (Other); Le Bonheur Children's Hospital (Other); Children's Hospital Colorado (Other); Nemours Children's Health System (Other); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Joseph Cravero, MD, Boston Children's Hospital
Other Study IDs: P00031812
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective is to create a multicenter registry which captures information relating to the perioperative anesthesia course and management of children undergoing anterior cruciate ligament reconstruction and to examine practice patterns and incidence of complications. Data from any single institution involved in this registry will be used for local safety and quality improvement efforts. In addition data from each institution can be compared to the information from the entire group of institutions participating in the project, thus providing a measure for comparison with national practice. The aggregate multi-institutional data set will be used to develop quality benchmarks for national safety and quality improvement efforts and best practice recommendation. We believe that this registry can also demonstrate how web based data collection can be used to evaluate clinical anesthesia outcomes for surgeries with a low incidence of critical events but with significant variability in medical management.

DETAILED DESCRIPTION:
This multi institutional registry will capture data relating to perioperative practices and complications, some of which may be relatively infrequent. The goal of this group is to create this registry to be used for local safety and quality improvement and multi-center benchmarking in this population. Reports generated from the registry will provide individual institutions with comparative data showing how their site performs compared to composite averages from all participating sites. Queries of the composite data set may allow for identification of factors associated with improved outcomes in this population. Future queries of the data-base for research purposes will require approval of the participating members of SPAIN.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 12 years to 17.5 years
* Patients undergoing scheduled surgical procedures on the anterior cruciate ligament construction surgery in a hospital setting or surgical day center.

Exclusion Criteria:

* Incarcerated subjects
* Non-English speaking families and subjects

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children undergoing scheduled surgical procedures on the anterior cruciate ligament in a hospital setting or surgical day center, aged 12-18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Registry Creation | 2 years
  The development of a multi-center registry of all anterior cruciate ligament reconstruction performed in the pediatric population with anterior cruciate ligament tear.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cravero, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Waltham, Massachusetts

REFERENCES:
- [Derived] Mandler T, Li G, Sadacharam K, Staffa SJ, Chidambaran V, O'Brien E, Kastner Ungar G, Muhly WT, Cravero J, Fernandez AM; SPAIN-ACL Investigators. Regional anesthesia and functional outcomes after anterior cruciate ligament reconstruction surgery in adolescent patients: Society of Pediatric Anesthesia Improvement Network (SPAIN). Reg Anesth Pain Med. 2025 Oct 29:rapm-2025-107017. doi: 10.1136/rapm-2025-107017. Online ahead of print. PMID 41167613
- [Derived] Sadacharam K, Mandler T, Staffa SJ, Pestieau SR, Fuller C, Ellington M, Sparks JW, Fernandez AM; SPAIN-ACL Investigators. Regional Anesthesia and Pain Outcomes After Anterior Cruciate Ligament Reconstruction Surgery in Pediatric Patients: Society of Pediatric Anesthesia Improvement Network. Anesth Analg. 2026 Jan 1;142(1):93-101. doi: 10.1213/ANE.0000000000007376. Epub 2025 Jan 29. PMID 39879136